CLINICAL TRIAL: NCT02192229
Title: Safety and Efficacy Evaluation of the Dose Regimen of Vitamin D 50,000 IU(Biodal) Tablet Supplementation in the Treatment of Population With Vitamin D Deficiency.
Brief Title: Efficacy of the Dose Regimen of Oral Vitamin D 50,000 IU in the Treatment of Vitamin D Deficiency
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hayat Pharmaceutical Co. PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1150-5248
Record Dates: First submitted 2013-12-23; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Active Comparator): The intervention group will be supplemented with 50.000 IU vitamin D3 every week for 12 consecutive weeks
  Interventions: Drug: 50.000 IU vitamin D3 (Biodal 50,000 IU)
- Placebo group (Placebo Comparator): The placebo group will receive placebo Tablet which will be manufactured in a pharmaceutical factory to be identical to vitamin D3 Tablet in color, shape, size, and packaging
  Interventions: Drug: Placebo (to mimic Biodal 50,000 IU)

INTERVENTIONS:
Drug: 50.000 IU vitamin D3 (Biodal 50,000 IU)
  Other Names: Biodal 50,000 IU
  Arms: intervention group
Drug: Placebo (to mimic Biodal 50,000 IU) — Placebo Tablet will be manufactured in a pharmaceutical factory to be identical to vitamin D3 Tablet in color, shape, size, and packaging
  Arms: Placebo group

SUMMARY:
Abstract:

The main objective of the proposed study is to examine the Safety and Efficacy Evaluation of the Dose Regimen of Vitamin D 50,000 IU (Biodal) tablet supplementation in the treatment of population with vitamin D deficiency.

A randomized, double-blind placebo, Parallel design comparing vitamin D with Placebo will be conducted on 60 Healthy males and females with vitamin D deficiency, age from 18 to 49 years who attend the rehabilitation clinics at Jordan University Hospital .Participants who met the inclusion criteria will be asked to sign an informed witnessed consent form. Results obtained are expected to assess the safety and efficacy of the dose regimen used in this study as per Biodal SmPC. This study will also contribute to the global body of knowledge in this field. The major findings generated from this study could open certain avenues for further research through the association of the status of vitamin D in serum .

DETAILED DESCRIPTION:
The study design will be a prospective randomized double blind parallel design comparing Vitamin D with Placebo. This study will be conducted in Jordan University Hospital (JUH). The participants will be Healthy males and females with vitamin D deficiency (18 to 49 years old). All eligible males and females who agree to participate in the study will sign an informed witnessed consent form at the beginning of the study. The expected duration of participants participation will be around 120 days and the number of visits for each participant will be 6 visits divided as follows; the first visit will be before 7 days of the initiation of the trial (screening period), the second on day zero of the treatment period, the third on day 30, the fourth on day 60, the fifth on day 90 and the sixth or the last visit will be on day 104 (after 14 days of the last treatment). Therefore the treatment period will be 90 days and the post treatment follow up period will be 14 days.

ELIGIBILITY:
Inclusion criteria:

* Subject is willing and able to give voluntary informed consent for participation in the study.
* Ethnic group (Caucasian).
* Healthy males or females aged between 18 and 49 years old.
* Normal weight (BMI 18.5-25kg/m2).
* Physical examination being assessed and accepted by the attending physician.
* Systolic blood pressure within the normal range (90-140) mmHg.
* Diastolic blood pressure within the normal range (60-90) mmHg.
* Heart rate within the normal range (60-100 beats/min).
* Oral body temperature within the normal range (35.9 - 37.6 Cº).
* Diagnosed with vitamin D deficiency with 25-OH Vitamin D level < 20ng/ml.
* All laboratory tests which including : Urine analysis, Hematology (Hb, Packed Cell Volume, Red Blood Cell, Mean Corpuscular Hemoglobin , Mean Corpuscular Hemoglobin Concentration , Mea Corpuscular Volume, Leukocytes, Lymphocytes, Eosinophils, Basophils, Monocytes, Neutrophils, Platelet count), Kidney function tests, Liver function test, Virology, Clinical chemistry, Ca, Mg, PO4, PTH , Alkaline Phosphatase and pregnancy test for married females ,results within the normal reference range.
* Able and willing to comply with all study requirements.

Exclusion Criteria

The subject may not enter the study if ANY of the following apply:

* Female subjects who is pregnant, lactating or planning pregnancy during the course of the study.
* Ethnic group non Caucasian.
* Males and Females aged <18 or >49 years old.
* Underweight, overweight and obese Females and males
* Males and Females diagnosed with diabetes, hypothyroidism, hyperthyroidism, liver disease, renal dysfunction, cardiovascular diseases including hypertension, androgen-secreting tumor, Cushing syndrome, congenital adrenal hyperplasia, hyperprolactinemia, and/or virilism.
* Known history or presence of food allergies or intolerance (e.g dairy products or gluten containing food), or any known condition that could interfere with the absorption, distribution, metabolism or execration of drugs.
* History of drug or alcohol abuse, smoking of 10 cigarettes or more (or equivalent) per day.
* Subjects who took medications known to affect metabolic parameters, such as metformin and corticosteroid drugs, vitamin D and calcium.
* Participation in another clinical or bioequivalence study within 90 days prior to the start of this study period.
* Subjects with abnormal ECG.
* Subjects with any abnormal laboratory results except 25 OH-Cholecalciferol level.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of the dose regimen considered in this study as the product SmPC which will be measured through the assessment of serum 25 (OH)D along the trial period. | 14 weeks
  To assess the dose regimen effectiveness used in this study as per Biodal SmPC.

SECONDARY OUTCOMES:
Assessing the level of (Urine analysis, Hematology ,Kidney Function Test,Liver Function Test, Virology, chemistry, 25(OH)D, Ca, Mg, Phosphate, Parathyroid hormone, Alkaline Phosphatase ) and reporting any adverse events through the trial period. | 14 weeks
  Evaluation of the safety of the dose regimen of vitamin D3 supplementation which will be measured by assessing the level of laboratory tests which including (Urine analysis Hematology Kidney function tests, Liver function test, Virology, Clinical chemistry, 25(OH)D, Ca, Mg, PO4, PTH , Alkaline Phosphatase and pregnancy test for married females), Physical examinations ,ECG examination, vital signs, and reporting any adverse events through the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Talal Aburjai, Ph.D., Principal Investigator — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan